CLINICAL TRIAL: NCT02380469
Title: Improvement of Information to Cancer Patients' Caregivers: a Randomised Intervention Study
Brief Title: Improvement of Information to Cancer Patients' Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Danish Cancer Society (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Mogens Groenvold, Professor, DMSc, PhD, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R82-A5445
Record Dates: First submitted 2015-01-29; First posted 2015-03-05 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Neoplasms
Keywords: Caregivers; Cancer; Information; Intervention; Randomised trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Experimental): Immediately after enrollment in the project, caregivers and patients receive the intervention
  Interventions: Behavioral: Identification and provision of lacking information
- Delayed intervention (3 weeks later) (Other): This group receives the same intervention as in the experimental group, but after the outcome assessment at 2 weeks
  Interventions: Behavioral: Identification and provision of lacking information

INTERVENTIONS:
Behavioral: Identification and provision of lacking information — The intervention consists of an interview about the caregiver's responses (baseline measurement) to a list about 'lack of information' within 13 areas. For each area, the patient's nurse will enquire about what information is requested by the caregiver and the patient. Subsequently, the nurse provides the requested information. She may involve the doctor and arrange follow-up visits or phone calls until the need is covered

SUMMARY:
The purpose of this study is to investigate whether a systematic early assessment of uncovered needs for information, supplemented by an interview about the needs with the patient's nurse who seeks to provide the information requested, will improve the caregivers' and the patients' satisfaction with information and communication and potentially also decrease anxiety and depression.

ELIGIBILITY:
Patient Inclusion Criteria:

* Cancer patient
* Newly refered to (i.e., this is the patient's first visit in) Department of Oncology, Herlev Hospital, in order to start medical treatment (e.g. chemotherapy)
* Written informed consent

Caregiver Inclusion Criteria:

* Attends the first visit in the Department of Oncology with the patient
* Has lacked information about at least one of the 13 aspects of information asked about in the questionnaire
* Written informed consent

Exclusion Criteria:

* Patient and/or caregiver do not understand Danish well enough to participate in the study
* The patient has an expected survival of less than six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Satisfaction with information from health care professionals | Change from baseline (enrollment) at 2 weeks
  Measure: The "Cancer Caregiving Tasks, Consequences and Needs Questionnaire" (CaTCoN) item 24

SECONDARY OUTCOMES:
Satisfaction with information from health care professionals | Change from baseline (enrollment) at 2 weeks
  Measure: CaTCoN subscale "Lack of information from health care professionals" (revised version)
Satisfaction with communication with health care professionals | Change from baseline (enrollment) at 2 weeks
  Measure: CaTCoN subscale "Problems with the quality of information and communication from health care professionals"
Satisfaction with support from health care professionals | Change from baseline (enrollment) at 2 weeks
  Measures: CaTCoN subscale "Lack of attention from health care professionals on the caregivers' wellbeing"
Satisfaction with support from health care professionals | Change from baseline (enrollment) at 2 weeks
  Measures: CaTCoN subscale "Need for help from health care professionals"
Anxiety and depression | Change from baseline (enrollment) at 2 weeks
  Measure: The Hospital Anxiety and Depression Scale (HADS)
Fulfillment of needs | Change from baseline (enrollment) at 2 weeks
  Measure: Family Inventory of Needs (FIN)

OTHER OUTCOMES:
The time spent on information as reported by health care professionals | Weeks 0-6 from baseline
  Investigated in focus group interviews with the health care professionals
Satisfaction with information from health care professionals | Change from baseline (enrollment) at 12 weeks
  Measure: CaTCoN item 24
Satisfaction with information from health care professionals | Change from baseline (enrollment) at 12 weeks
  Measure: CaTCoN subscale "Lack of information from health care professionals" (revised version)
Satisfaction with communication with health care professionals | Change from baseline (enrollment) at 12 weeks
  Measure: CaTCoN subscale "Problems with the quality of information and communication from health care professionals"
Satisfaction with support from health care professionals | Change from baseline (enrollment) at 12 weeks
  Measures: CaTCoN subscale "Lack of attention from health care professionals on the caregivers' wellbeing"
Satisfaction with support from health care professionals | Change from baseline (enrollment) at 12 weeks
  Measures: CaTCoN subscale "Need for help from health care professionals"
Anxiety and depression | Change from baseline (enrollment) at 12 weeks
  Measure: The Hospital Anxiety and Depression Scale (HADS)
Fulfillment of needs | Change from baseline (enrollment) at 12 weeks
  Measure: Family Inventory of Needs (FIN)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Groenvold, DMSc PhD MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Oncology, Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Background] Lund L, Ross L, Groenvold M. The initial development of the 'Cancer Caregiving Tasks, Consequences and Needs Questionnaire' (CaTCoN). Acta Oncol. 2012 Nov;51(8):1009-19. doi: 10.3109/0284186X.2012.681697. Epub 2012 May 8. PMID 22564144
- [Background] Lund L, Ross L, Petersen MA, Groenvold M. The validity and reliability of the 'Cancer Caregiving Tasks, Consequences and Needs Questionnaire' (CaTCoN). Acta Oncol. 2014 Jul;53(7):966-74. doi: 10.3109/0284186X.2014.888496. Epub 2014 Mar 16. PMID 24628263
- [Background] Lund L, Ross L, Petersen MA, Groenvold M. The interaction between informal cancer caregivers and health care professionals: a survey of caregivers' experiences of problems and unmet needs. Support Care Cancer. 2015 Jun;23(6):1719-33. doi: 10.1007/s00520-014-2529-0. Epub 2014 Nov 29. PMID 25432867
- [Derived] Lund L, Ross L, Petersen MA, Sengelov L, Groenvold M. Improving information to caregivers of cancer patients: the Herlev Hospital Empowerment of Relatives through More and Earlier information Supply (HERMES) randomized controlled trial. Support Care Cancer. 2020 Feb;28(2):939-950. doi: 10.1007/s00520-019-04900-3. Epub 2019 Jun 8. PMID 31177391